CLINICAL TRIAL: NCT01126619
Title: To Observe the Effectiveness and Safety of Anti-TNFs in Patients With Moderate to Severe Psoriasis
Brief Title: A Study of Effectiveness and Safety of Tumor Necrosis Factor (TNF) Inhibitors in Patients With Moderate to Severe Psoriasis
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: P12-130
Record Dates: First submitted 2010-05-18; First posted 2010-05-20 (Estimated); Results first posted 2012-10-11 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: Psoriasis
Keywords: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- Anti-TNF: Participants with moderate to severe psoriasis who were prescribed an Anti Tumor Necrosis Factor (anti-TNF) agent prior to enrollment according to national approved indications and reimbursement guidelines.

SUMMARY:
In recent years, biologics have changed the treatment of psoriasis, giving us additional therapeutic options that are potentially less toxic to the liver, kidneys, and bone marrow and are not teratogenic. Nevertheless, traditional systemic therapies continue to play an important role in the treatment of psoriasis in Turkey, even in patients who are requiring biologic treatments according to national recommendations. This study is designated to observe the effectiveness and safety of tumor necrosis factor inhibitors in patients with moderate to severe psoriasis.

DETAILED DESCRIPTION:
Patients admitted to dermatology clinics, with moderate to severe psoriasis for whom the physician has decided to initiate psoriasis treatment with anti-TNFs in accordance with Turkish Ministry of Health regulations and reimbursements. (Tumor necrosis factor inhibitors can be used for the treatment of moderate to severe chronic plaque psoriasis in adult patients who failed to respond to or who have a contraindication to, or are intolerant to other systemic therapy including cyclosporine, methotrexate or Psoralen Ultra-Violet A. Patients should be screened for latent tuberculosis and appropriate anti-tuberculosis prophylaxis must be initiated if latent tuberculosis is diagnosed). This is a national, multi-center, observational, prospective photographic atlas study in patients who are treated with tumor necrosis factor inhibitors for moderate to severe psoriasis in daily clinic according to Turkish regulations and reimbursement. Demographic data will be collected by the investigator at the beginning of the study. Every participant will be examined by the investigator and the Psoriasis Area Severity Index will be determined at the beginning of the study and at weeks 4, 8, 16 and 24. Each patient will be asked to fill out the Dermatology Life Quality Index at each visit. Each patient will be asked to fill out the Work Productivity and Activity Impairment Questionnaire: Psoriasis at the beginning and last visit (week 24). A standardized set of photographs will be taken at the beginning of the study and at weeks 4, 8, 16 and 24 by a dermatologist trained about standardized photograph positioning and settings. Psoriasis Area Severity Index, Dermatology Life Quality Index and Photographic scores will be statistically analyzed separately in order to evaluate treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥18 years old with moderate-to-severe psoriasis.
* Patients for whom the physician has decided to initiate psoriasis treatment with anti-TNFs in accordance with Turkish Ministry of Health regulations and reimbursements.
* Patients who are able to understand and answer a self administered questionnaire.
* Patients signed an informed consent form stating that they agreed to have their photographs taken, analyzed, and included in a scientific publication.

Exclusion Criteria:

* Patients who do not consent to being photographed during the study.
* Females who are pregnant, nursing, or of childbearing potential who refuse to use a medically acceptable form of contraception throughout the study.
* Patients with untreated tuberculosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: University hospitals in Turkey
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2010-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mahmut Gucuk, MD, Study Director — Abbott Laboratories Ithalat, Ithalat ve Tic. Ltd. Sti
Locations (25):
- Turkey (Türkiye) (25):
  - Site Reference ID/Investigator# 38780, Afyonkarahisar
  - Site Reference ID/Investigator# 27422, Ankara
  - Site Reference ID/Investigator# 38776, Ankara
  - Site Reference ID/Investigator# 38777, Ankara
  - Site Reference ID/Investigator# 38763, Ankara
  - Site Reference ID/Investigator# 38767, Aydin
  - Site Reference ID/Investigator# 38769, Bursa
  - Site Reference ID/Investigator# 38779, Edirne
  - Site Reference ID/Investigator# 38782, Gaziantep
  - Site Reference ID/Investigator# 38778, Hatay
  - Site Reference ID/Investigator# 38786, Isparta
  - Site Reference ID/Investigator# 38765, Istanbul
  - Site Reference ID/Investigator# 38771, Istanbul
  - Site Reference ID/Investigator# 38766, Istanbul
  - Site Reference ID/Investigator# 38770, Istanbul
  - Site Reference ID/Investigator# 38764, Izmir
  - Site Reference ID/Investigator# 44104, Kocaeli
  - Site Reference ID/Investigator# 38781, Konya
  - Site Reference ID/Investigator# 44102, Kırıkkale
  - Site Reference ID/Investigator# 38773, Malatya
  - Site Reference ID/Investigator# 38768, Manisa
  - Site Reference ID/Investigator# 38772, Mersin
  - Site Reference ID/Investigator# 44262, Samsun
  - Site Reference ID/Investigator# 44103, Sivas
  - Site Reference ID/Investigator# 44105, Zonguldak

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anti-TNF
Started | 103
Completed | 86 (The completed population was used for all effectiveness analyses.)
Not Completed | 17
Not completed — Not eligible for the study | 2
Not completed — Investigator decision | 4
Not completed — Serious adverse event | 1
Not completed — Withdrawal by Subject | 9
Not completed — Non-compliance | 1

BASELINE CHARACTERISTICS:
Arm/Group | Anti-TNF
Number analyzed (Participants) | 103
Age Continuous [Mean (Standard Deviation); unit: years] — Data available for 102 participants.
  years | 44.9 (13.9)
Gender [Number; unit: participants] — Data available for 102 participants.
  participants
    Female | 40
    Male | 62
Region of Enrollment [Number; unit: participants]
  Turkey | 103
Weight [Mean (Standard Deviation); unit: kg] — Data available for 102 participants.
  kg | 78.5 (16.0)
Height [Mean (Standard Deviation); unit: cm] — Data available for 101 participants.
  cm | 166.9 (13.5)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Data available for 101 participants.
  kg/m^2 | 29.3 (14.9)
Psoriasis Area and Severity Index (PASI) Score [Mean (Standard Deviation); unit: scores on a scale] — Psoriasis Area and Severity Index (PASI) score is based on assessment of erythema (reddening), induration (plaque thickness), desquamation (scaling), and area affected as observed on the day of examination. The score ranges from 0 (best outcome) to 72 (worst outcome).
  scores on a scale | 20.8 (11.2)
Dermatology Life Quality Index (DLQI) Score [Mean (Standard Deviation); unit: scores on a scale] — DLQI is a questionnaire to evaluate dermatology patients for their quality of life for the following subsets of parameters: symptoms and feelings, daily activities, leisure activities, work or school activities, personal relationships and treatment related feelings. Questions related with these parameters are summed up and the range of the total score is 0 to 30. A score of 21 to 30 means an extremely large effect on patient's life whereas 0-1 means that the disease has no effect at all.
  scores on a scale | 15.1 (7.3)
Duration of Psoriasis [Mean (Standard Deviation); unit: years] — Data available for 102 participants.
  years | 15.7 (9.2)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Psoriasis Area and Severity Index (PASI) Score
Description: The Psoriasis Area and Severity Index (PASI) score is a combination of the intensity of psoriasis, assessed by the erythema (reddening), induration (plaque thickness) and desquamation (scaling) on a scale from none (0), mild (1), moderate (2), severe (3) or very severe (4), together with the percentage of the area affected, rated on a scale from 0 to 6. PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 to 72. The higher the total score, the more severe the disease. Change from Baseline is presented as a percentage of the Baseline value: Baseline value - post-baseline value / Baseline value * 100.
Time Frame: Baseline and Weeks 4, 8, 16 and 24
Population: Participants who received treatment with anti-TNF agents and completed study follow-up visits through to Week 24.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Anti-TNF
Number analyzed (Participants) | 86
Percent change
  Week 4 | 48.65 (36.27)
  Week 8 | 75.70 (36.11)
  Week 16 | 87.85 (36.91)
  Week 24 | 90.29 (25.49)

2. Secondary Outcome: Dynamic Physician Global Assessment (PGA) of Change in Psoriasis
Description: In the dynamic physician global assessment of change in psoriasis, the physician compared sets of standardized photographs taken at Baseline and at Week 24 for each participant and rated the change of psoriasis severity on the dynamic PGA scale from -5 (considerable deterioration), 0 (no or minimal change) to +5 (considerable improvement).
Time Frame: Baseline and Week 24
Population: Participants who received treatment with anti-TNF agents and completed study follow-up visits through to Week 24.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Anti-TNF
Number analyzed (Participants) | 86
scores on a scale | 1.51 (2.24)

3. Secondary Outcome: Dynamic Patient Global Assessment (PGA) of Change in Psoriasis
Description: In the dynamic patient global assessment of change in psoriasis, the participant compared their own sets of standardized photographs taken at Baseline and at Week 24 and rated the change of the severity of psoriasis using the dynamic photographic scale adapted to a visual analog scale ranging from -5 (very large deterioration) to +5 (very large improvement).
Time Frame: Baseline and Week 24
Population: Participants who received treatment with anti-TNF agents and completed study follow-up visits through to Week 24.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Anti-TNF
Number analyzed (Participants) | 86
scores on a scale | 1.51 (2.26)

4. Secondary Outcome: Static Physician Global Assessment (PGA) of Psoriasis
Description: In the static physician assessment of psoriasis, psoriasis severity was rated first for all Baseline photographs and then for all Week 24 photographs according to the following scale:
  Clear (no lesion); Psoriasis almost cleared; Mild psoriasis; Mild to moderate psoriasis; Moderate psoriasis; Moderate to severe psoriasis; Severe psoriasis.
Time Frame: Baseline and Week 24
Population: Participants who received treatment with anti-TNF agents and completed study follow-up visits through to Week 24.
Measure: Number; unit: participants
Groups:
- Baseline: Baseline Static Physician Global Assessment of Psoriasis, prior to initiation of anti-TNF therapy.
- Week 24: Week 24 Static Physician Global Assessment of Psoriasis, after 24 weeks of anti-TNF therapy.
Arm/Group | Baseline | Week 24
Number analyzed (Participants) | 86 | 86
participants
  Clear psoriasis | 0 | 14
  Psoriasis almost clear | 0 | 38
  Mild psoriasis | 0 | 19
  Mild to moderate psoriasis | 1 | 4
  Moderate psoriasis | 35 | 8
  Moderate to severe psoriasis | 27 | 3
  Severe psoriasis | 23 | 0

5. Secondary Outcome: Percent Change From Baseline in Dermatology Life Quality Index (DLQI) Score
Description: The DLQI questionnaire asks participants to evaluate the degree that psoriasis has affected their quality of life in the last week, and includes the following parameters: symptoms and feelings, daily activities, leisure activities, work or school activities, personal relationships and treatment related feelings. Participants answer 10 questions on a scale from 0 (not at all) to 3 (very much); the range of the total score is 0 to 30. A score of 21 to 30 means an extremely large effect on the participant's life whereas 0-1 means that the disease has no effect at all.
  Change from Baseline is presented as a percentage of the Baseline value: Baseline value - post-baseline value / Baseline value * 100.
Time Frame: Baseline and Weeks 4, 8, 16 and 24
Population: Participants who received treatment with anti-TNF agents and completed study follow-up visits through to Week 24.
Measure: Mean (Full Range); unit: percent change
Arm/Group | Anti-TNF
Number analyzed (Participants) | 86
percent change
  Week 4 | 53.13 [-133.33 to 100.00]
  Week 8 | 66.40 [-80.00 to 100.00]
  Week 16 | 73.98 [-58.33 to 100.00]
  Week 24 | 65.72 [-166.67 to 100.00]

6. Primary Outcome: Percentage of Participants With 75% Reduction in PASI Score
Description: The percentage of participants with a 75% reduction (improvement) in Psoriasis Area and Severity Index (PASI) score from Baseline. PASI score is based on an assessment of erythema (reddening), induration (plaque thickness), desquamation (scaling), and the percent area affected as observed on the day of examination. The score ranges from 0 (best outcome) to 72 (worst outcome).
Time Frame: Baseline and Weeks 4, 8, 16 and 24
Population: Participants who received treatment with anti-TNF agents and completed study follow-up visits through to Week 24.
Measure: Number; unit: percentage of participants
Arm/Group | Anti-TNF
Number analyzed (Participants) | 86
percentage of participants
  Week 4 | 31.4
  Week 8 | 51.2
  Week 16 | 67.4
  Week 24 | 70.9

7. Secondary Outcome: Percent Change From Baseline in Work Productivity and Activity Impairment
Description: The following parameters were assessed using the Work Productivity and Activity Impairment Questionnaire: Psoriasis (WPAI:PSO):
  * Percent work time missed in the last 7 days due to problems associated with psoriasis;
  * Percent impairment at work, based on the participant's assessment of how much psoriasis affected their productivity while they were working in the last 7 days;
  * Percent overall loss of work productivity, based on hours missed and impairment while working due to psoriasis;
  * Percent general activity impairment, based on the participant's assessment of how much psoriasis affected their ability to perform regular daily activities, such as work around the house, shopping, child care, exercising, studying, etc.
  Each domain score ranges from 0 (no impairment) to 100 (complete impairment). Change from Baseline is presented as a percentage of the Baseline value: Baseline value - post-baseline value / Baseline value * 100.
Time Frame: Baseline and Week 24
Population: Participants who received treatment with anti-TNF agents and completed study follow-up visits through to Week 24. The first 3 domains (work time missed, work impairment and overall loss of work productivity) were assessed on a sub-group of participants who had full time jobs (n=30).
Measure: Mean (Full Range); unit: percent change
Arm/Group | Anti-TNF
Number analyzed (Participants) | 86
percent change
  Work time missed | 96 [0 to 100]
  Impairment at work | 72 [0 to 100]
  Overall loss of work productivity | 75 [0 to 100]
  Activity impairment | 72 [0 to 100]

8. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: The number of participants experiencing any adverse event or a serious adverse event during the study are summarized. A serious AE is an event that results in death, is life-threatening, requires or prolongs hospitalization, is a congenital anomaly, results in persistent or significant disability/incapacity or is an important medical event that may require medical or surgical intervention to prevent any of the outcomes listed above.
  Please see the Adverse Event module below for additional details.
Time Frame: 24 Weeks
Population: All enrolled participants.
Measure: Number; unit: participants
Arm/Group | Anti-TNF
Number analyzed (Participants) | 103
participants
  Any adverse event | 28
  Serious adverse event | 3

ADVERSE EVENTS:
Time Frame: 24 weeks.
Arm/Group | Anti-TNF
Serious Adverse Events (participants affected / at risk) | 3/103
Other Adverse Events (participants affected / at risk) | 7/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anti-TNF (N=103)
Hepatotoxicity, Toxic Hepatitis (Gastrointestinal disorders) | 1
Gangrenous emphysema (Respiratory, thoracic and mediastinal disorders) | 1
Catheter infection, infected endocarditis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Anti-TNF (N=103)
Injection site reaction (General disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.